CLINICAL TRIAL: NCT04449471
Title: Project 1: Program on Genetic and Dietary Predictors of Drug Response in Rural and AI/AN Populations (Naproxen Study)
Brief Title: Naproxen Pharmacogenetic Study (Project 1, Aim 2)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Oregon Health and Science University (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Kenneth Thummel, Professor: Pharmaceutics, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SITE00000671; 5P01GM116691 (NIH)
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Pharmacogenetics
Keywords: CYP2C9; naproxen; polymorphism
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Intervention Model Description: Healthy adults with predetermined CYP2C9 genotype will receive the probe drug, naproxen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Naproxen Tablet (Experimental): Subjects will received a single 220-mg dose of naproxen sodium (Aleve) by mouth.
  Interventions: Drug: Naproxen tablet

INTERVENTIONS:
Drug: Naproxen tablet — For this single intervention arm, each subject will receive a single 220-mg dose of naproxen sodium (Aleve), followed by urine collection for 24-hours.
  Other Names: Aleve

SUMMARY:
This is a mechanism-based study in healthy adults to determine the effect of the CYP2C9 M1L gene polymorphism on the functional activity of the encoded CYP2C9 enzyme towards the probe substrate naproxen. CYP2C9 activity will be evaluated by measurement of O-desmethyl naproxen and unchanged naproxen in 24-hour urine following administration of a single oral dose of naproxen (Aleve) in Yup'ik Alaska Native adult men and women who were previously determined in a separate observational study to be homozygous for the CYP2C9*1 allele or a carrier of the CYP2C9 M1L allele.

DETAILED DESCRIPTION:
This pharmacogenetics study will test the hypothesis that inheritance of a M1L variant in the CYP2C9 gene, which was first discovered in Yup'ik Alaska Native people, causes complete loss of function in CYP-2C9-dependent catalytic activity.

Study participants will be selected from a cross-sectional population of >750 Yup'ik men and women, ≥18 years, for whom CYP2C9 genotype has already been determined as part of a SNP discovery study, and who consented to be contacted for future research. There will be 15 participants in each of two genotyped groups ((1) Met1/Met1 and (2) Met1/Leu1 or Leu1/Leu1), for a total of 30 participants. The two groups will be matched for sex of the participants; the proportion determined by the composition of the least frequent Leu1 carrier group. The investigators will attempt to recruit a similar range of ages in each genotyped group and the widest range possible. Recruitment will occur in one of 10 communities in the Yukon-Kuskokwim delta that participated in our original SNP discovery study.

Participants will be asked to fast overnight prior to the study and will be allowed to eat ad libitum 2 hours after naproxen is taken. A fasting 13 ml venous blood sample will be collected from each participant for isolation of DNA and plasma. Spot urine will be collected from each participant as an analytic control the morning of the blood draw. At approximately 9 am, each participant will be given a single 220-mg dose of Naproxen, by mouth, with a glass of water. The total urine output over the next 24-hour will be collected by the participant and returned to the clinic the next day. The urine volume will be measured and recorded and two 5 mL aliquots will be frozen at -80°C and stored for unchanged drug and metabolite analysis analyses.

Total (conjugated and unconjugated) 6-O-Desmethyl naproxen and unchanged naproxen concentrations in urine will be measured by LC-MS/MS. A ratio of the total 6-O-desmethyl naproxen/naproxen (M/P) excreted in urine over 24-hours will be computed. 6-O-desmethyl naproxen is formed selectively by CYP2C9.

Pairwise comparison of the mean M/P ratios, assuming unequal variance, will be evaluated using a t-test to determine if there are significant differences in activity for carriers of the Leu 1 variant. The sample size provides 80% power to detect a difference, at a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. No history of significant medical conditions including cardiac, pulmonary, gastrointestinal, or renal disease, HIV, or history of asthma, urticaria, or allergic-type reactions with aspirin (ASA) or other NSAID (nonsteroidal anti-inflammatory drug).
2. Both males or females 18 years and older.
3. Self-identified as Yup'ik or Cup'ik
4. Able to read and understand English or Yup'ik.
5. Able to provide informed consent.
6. Women not currently pregnant or lactating.

Exclusion Criteria:

1. Individuals with any significant chronic medical condition, including cardiac, pulmonary, hepatic, gastrointestinal, or renal disease, HIV, or history of asthma, urticaria, or allergic-type reactions with aspirin (ASA) or other NSAID
2. Individuals less than 18 years of age.
3. Individuals unable to read and understand English or Yup'ik.
4. Individuals unable to provide informed consent.
5. Individuals taking drugs or natural products known to affect the metabolic activity of CYP2C9 (e.g., rifampin, carbamazepine, barbiturates, phenytoin, valproic acid, fluconazole, ketoconazole, miconazole, amiodarone, fluvastatin and milk thistle.
6. Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01-12 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
6-O-desmethyl naproxen/naproxen ratio | 24-hours
  A ratio of the total mount of 6-O-desmethyl naproxen/unchanged naproxen in 24-hour urine

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E. Thummel, PhD, Principal Investigator — University of Washington
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States